CLINICAL TRIAL: NCT01826240
Title: Mindfulness-Based Cognitive Therapy + Safety Planning For Suicidal Behavior: A Treatment Development Study
Brief Title: Mindfulness-Based Cognitive Therapy + Safety Planning For Suicidal Behavior
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6592; PDF-0-076-11 (Other Grant/Funding Number: American Foundation for Suicide Prevention)
Record Dates: First submitted 2013-03-13; First posted 2013-04-08 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2013-04

CONDITIONS: Monopolar Depression, Single Episode or Unspecified; Suicidal and Self-injurious Behaviour
MeSH Terms: conditions — Depression; Self-Injurious Behavior | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MBCT+SPI (Experimental): Note: There is only one condition in this study. Mindfulness-Based Cognitive Therapy (MBCT) is combined with Safety Planning Intervention (SPI). All individuals who choose to participate will receive MBCT+SPI.
  Interventions: Behavioral: MBCT+SPI

INTERVENTIONS:
Behavioral: MBCT+SPI — Safety Planning Intervention (SPI), a very brief intervention focused on identifying personalized coping strategies to manage acute suicidality, is combined with Mindfulness-Based Cognitive Therapy (MBCT), a group intervention comprised of mindfulness training and cognitive therapy techniques. Treatment lasts 9 weeks.
  Other Names: Mindfulness-Based Cognitive Therapy; Safety Planning Intervention

SUMMARY:
The purpose of this study is to combine and adapt Mindfulness-Based Cognitive Therapy (MBCT) + Safety Planning Intervention (SPI) for individuals with suicidal behavior and to determine its feasibility, acceptability, safety and preliminary effectiveness. An exploratory aim is to collect data on the cognitive changes underlying treatment gains.

DETAILED DESCRIPTION:
* The study is a nine-week clinical trial combining Safety Planning Intervention plus Mindfulness-Based Cognitive Therapy for patients with a recent history of suicidal thoughts or behavior and current or past depressive symptoms.
* These treatments work for depression and some preliminary data suggest they may work to prevent suicidal behavior.
* Participation includes:

  * Nine weeks of free treatment
  * Clinical assessments
  * An opportunity to offer your views on treatment and suggestions for improving the treatment in focus groups

ELIGIBILITY:
Inclusion Criteria:

* 18-65
* History of depression
* Suicidal behavior or thoughts (i.e., current suicidal thoughts at screening and history of at least one suicide attempt or suicide-related behavior (aborted or interrupted suicide attempt) or suicidal ideation with plan or method in the past 6 months)
* In active treatment (e.g., receiving psychiatric medications)

Exclusion Criteria:

* Current mania, psychosis, Obsessive-Compulsive Disorder, Traumatic Brain Damage, Organic or Acute Brain Syndrome, Mental Retardation or pervasive developmental disorder
* Requires priority treatment for an acute illness or debilitating problem such as severe primary substance dependence or anorexia nervosa
* Inability to complete psychiatric interview or group treatment due to lack of cooperation or lack of comprehension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Retention | participants will be followed for the duration of treatment, an expected average of 9 weeks
  Feasibility
Consumer Satisfaction Questionnaire | post-treatment (at 9 weeks)
  Acceptability
Change in scores on Scale for Suicide Ideation | participants will be followed for the duration of treatment, an expected average of 9 weeks
  Safety

SECONDARY OUTCOMES:
Change in scores on Beck Depression Inventory (BDI-II) | baseline and post-treatment (at 9 weeks)
  Effectiveness

OTHER OUTCOMES:
Change in cognitive processes underlying treatment gains | baseline and post-treatment (at 9 weeks)
  neuropsychological tasks assessing attention and other cognitive processes

CONTACTS AND LOCATIONS:
Overall Officials: Megan Chesin, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University/New York State Psychiatric Institute, New York, New York, United States